CLINICAL TRIAL: NCT00523757
Title: Aldosterone-blockade Randomized Controlled Trial In CHF - Diastolic
Brief Title: Aldosterone Blockade in Heart Failure
Acronym: ARCTIC-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Justin Ezekowitz (Other)
Responsible Party: Sponsor-Investigator, Justin Ezekowitz, Professor, University of Alberta
Organization: University of Alberta (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHF-G533000207
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: heart failure; collagen; diastolic function
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Spironolactone
  Interventions: Drug: Spironolactone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Heart failure causes significant morbidity and mortality and is the most rapidly increasing cardiovascular diagnosis in North America overall prevalence is estimated at 0.4% to 2.4%. Recently, heart failure with a preserved ejection fraction (HFNEF) was found in up to 50% of patients with symptomatic heart failure. Many studies have demonstrated that HFNEF has a poor prognosis with a mortality rate of up to 8% per year and a 50% chance of needing to be admitted to hospital in the next year. There are no proven therapies for this type of heart failure.

Aldosterone blockers (these drugs block a hormone that is elevated in patients with heart failure) are used in other types of heart failure. Our goal is to see if this type of drug improves the function of the heart by looking at the thickness of the heart muscle using MRI. Also we will measure the amount of tissue formation and breakdown in the heart. The trial will be done using both the drug and a placebo so that we can see what effects are due to the drug.

DETAILED DESCRIPTION:
Aldosterone antagonists have shown efficacy in systolic heart failure and in patients with post-myocardial infarction systolic dysfunction in three major randomized placebo controlled trials. Together these trials have demonstrated a reduction in mortality, hospitalization and a regression in left ventricular mass by MRI.

Primary Objective The primary objective of this study will be to assess the change in markers of collagen turnover and correlate this with specific measures of left ventricular mass regression and diastolic function on MRI after 4 months of aldosterone blockade.

Study Design and Methods This study is a double-blind, concealed allocation, randomized trial at the University of Alberta where patients with diastolic heart failure will be randomized to spironolactone or matching placebo for 4 months. Outcomes assessed include LV mass by MRI, collagen markers, other biomarkers, clinical outcomes, quality of life and exercise testing

ELIGIBILITY:
Inclusion Criteria:

1. HF by Framingham criteria
2. At least one admission to hospital for HF within the last 180 days
3. New York Heart Association Class II thru IV
4. Echocardiographic criteria:At least moderate diastolic dysfunction, Ejection fraction >45%

Exclusion Criteria:

1. Creatinine clearance <40 mls/min/1.73m2
2. Potassium >5.0 mmol/L
3. Recent acute coronary syndrome in the prior 4 weeks
4. Planned revascularization, defibrillator or pacemaker in next 4 months
5. Known previous intolerance to aldosterone antagonist

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04-30 (Actual); Study Completion 2010-04-30 (Actual)

PRIMARY OUTCOMES:
LVH | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ezekowitz, MBBCh MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada